CLINICAL TRIAL: NCT06320951
Title: Improving Cardiometabolic Health in Black Individuals Through Therapeutic Augmentation of Cyclic Guanosine Mono-Phosphate Signaling Pathway
Brief Title: VITAL-IMPACT: Improving Cardiometabolic Health in Black Individuals Through Therapeutic Augmentation of Cyclic Guanosine Mono-Phosphate Signaling Pathway
Acronym: VITAL-IMPACT
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Pankaj Arora, MD, Associate Professor, Division of Cardiovasular Disease, Department of Medicine, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 300012681; Pending (Other: Pending)
Record Dates: First submitted 2024-03-13; First posted 2024-03-20 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Cardiovascular Diseases; Insulin Sensitivity/Resistance; Metabolic Disease; Metabolism; Energy Expenditure; Obesity
Keywords: Energy Expenditure; Insulin Sensitivity; African Americans; Cyclic Guanosine Monophosphate
MeSH Terms: conditions — Cardiovascular Diseases; Insulin Resistance; Metabolic Diseases; Obesity | interventions — vericiguat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental: Vericiguat (Experimental): The subject will be randomized, in a double-blind manner to vericiguat 10 mg once daily for a period of 12 weeks.
  Interventions: Drug: Vericiguat 10 MG; Other: Insulin Sensitivity Test; Other: Resting Energy and Exercise Energy Expenditure Assessment; Other: White Adipose Tissue Biopsy; Other: MRI-PET Scan for Brown Adipose Tissue Volume Assessment
- Placebo (Placebo Comparator): The subject will be randomized, in a double-blind manner to placebo once daily for a period of 12 weeks.
  Interventions: Other: Placebo; Other: Insulin Sensitivity Test; Other: Resting Energy and Exercise Energy Expenditure Assessment; Other: White Adipose Tissue Biopsy; Other: MRI-PET Scan for Brown Adipose Tissue Volume Assessment

INTERVENTIONS:
Drug: Vericiguat 10 MG — The subject will be randomized, in a double-blind manner to vericiguat 10 mg once daily for a period of 12 weeks.
  Other Names: Vericiguat Arm
  Arms: Experimental: Vericiguat
Other: Placebo — The subject will be randomized, in a double-blind manner to placebo once daily for a period of 12 weeks.
  Other Names: Placebo Arm
  Arms: Placebo
Other: Insulin Sensitivity Test — An assessment of the insulin sensitivity will be done using the Euglycemic Hyperinsulinemic Clamp, at baseline and after 12 weeks of pharmacological interventions.
Other: Resting Energy and Exercise Energy Expenditure Assessment — Each participant's Energy Expenditure will be determined using a metabolic cart, at baseline and after 12 weeks of pharmacological interventions.
  Other Names: Resting and Exercise Induced Energy Expenditure Test
Other: White Adipose Tissue Biopsy — Participants who consent to participate in the exploratory aim will undergo WAT biopsy to assess UCP1 gene expression from the collected biospecimens, at baseline and after 12 weeks of pharmacological interventions.
Other: MRI-PET Scan for Brown Adipose Tissue Volume Assessment — Participants who consent to participate in the exploratory aim will undergo PET/MR to BAT volume at baseline and after 12 weeks of pharmacological interventions.

SUMMARY:
This study investigates the potential of vericiguat, a soluble guanylate cyclase stimulator, to improve cardiometabolic health in obese Black individuals with insulin resistance by directly enhancing cyclic guanosine monophosphate (cGMP) activity. Given that this population has been shown to have lower cGMP activity and the association of lower cGMP activity with increased cardiometabolic disease risk, the proposed study hypothesizes that augmenting cGMP activity in obese individuals will improve insulin sensitivity and energy expenditure. This study is a placebo-controlled randomized trial involving 200 Black obese participants with insulin resistance, assessing the effects of vericiguat on insulin sensitivity, resting, and exercise-induced energy expenditure over 12 weeks. Additionally, it will explore changes in brown adipose tissue and gene expression related to energy metabolism in white adipose tissue, aiming to provide insights into how increasing cGMP activity may improve cardiometabolic health in Black obese individuals.

DETAILED DESCRIPTION:
Obese Black individuals have a higher prevalence of insulin resistance, which is linked to an elevated risk of cardiometabolic diseases and cardiovascular disease. The reasons behind the increased insulin resistance in this group are not fully understood. Key to regulating glucose metabolism and the overall balance of energy, the cyclic guanosine monophosphate (cGMP) pathway is crucial for maintaining cardiometabolic health. Research indicates that both Black race and obesity are associated with reduced levels of upstream regulators of cGMP activity, including natriuretic peptides (NPs) and nitric oxide (NO). This reduced level of NPs and NO predisposes Black obese individuals to decreased cGMP activity, potentially contributing to the higher occurrence of cardiometabolic diseases seen in this population. Vericiguat, a drug that stimulates the soluble guanylate cyclase, thereby enhancing cGMP activity independently of NO, presents a novel approach to improving cardiometabolic health in those most at risk due to low cGMP activity. This study hypothesizes that directly augmenting cGMP levels with vericiguat will improve cardiometabolic health parameters including insulin sensitivity and energy expenditure in Black obese adults with insulin resistance. Investigators plan to execute a placebo-controlled randomized trial targeting Black obese participants with insulin resistance to examine whether vericiguat can (1) improve insulin sensitivity and (2) increase resting energy expenditure. For the first aim, Investigators aim to enroll 200 Black obese (BMI≥30 kg/m^2) individuals with a HOMA-IR of ≥2.5, randomizing them to either vericiguat 10 mg once daily or a placebo once daily in a double-blind setup for 12 weeks. Investigators will assess improvements in insulin sensitivity through euglycemic hyperinsulinemic clamp and compare the results between the vericiguat and placebo groups after 12 weeks. For the second aim, Investigators will evaluate changes in resting and exercise energy expenditure across both groups over the same period. An exploratory objective will investigate changes in brown adipose tissue volume and activity using PET-MRI, as well as UCP1 gene expression in white adipose tissue, in a subset of 100 participants after 12 weeks of vericiguat treatment. This will offer insights into the mechanisms by which cGMP augmentation may facilitate improvements in cardiometabolic health. By focusing on the direct enhancement of cGMP activity in Black obese individuals, this study proposes a novel targeted therapeutic strategy aimed at improving cardiometabolic health and addressing the increasing prevalence of cardiometabolic disease in the Black population.

ELIGIBILITY:
Inclusion Criteria:

* Adults: Age more than or equal to 18 years of age
* Self-identified race/ethnicity as African-American or Black
* BMI ≥ 30 kg/m2
* HOMA-IR ≥ 2.5
* Blood pressure: 120-160/80-100 mmHg (untreated or 1 week of washout in those treated with up to two classes of antihypertensives)
* Willing to adhere to study protocol

Exclusion Criteria:

* Women who are pregnant or breastfeeding or who can become pregnant and not practicing an acceptable method of birth control during the study (including abstinence)
* Have any past or present history of cardiovascular diseases (stroke, myocardial infarction, heart failure, transient ischemic attack, angina, seizure or cardiac arrhythmia)
* BP more than 160/100 mmHg or those treated with three or more classes of antihypertensives
* BMI >45 kg/m2
* History of diabetes or fasting plasma glucose >=126 mg/dL or HbA1C>=6.5% or prior treatment with antidiabetics
* Estimated GFR < 60 ml/min/1.73 m2; albumin-creatinine ratio ≥30 mg/g
* Hepatic Transaminase (AST and ALT) levels >3x the upper limit of normal
* Significant psychiatric illness (assessed using validated MINI questionnaire)
* Anemia (men, Hb<13 g/dL; women, Hb <12 g/dL)
* Inability to exercise on a treadmill

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-12-01 (Estimated); Primary Completion 2028-04-30 (Estimated); Study Completion 2029-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in insulin sensitivity after vericiguat in Black obese individuals with insulin resistance. | 12 weeks
  The difference in change in insulin sensitivity between baseline and post-intervention between two arms.
Change in resting energy expenditure (REE) after vericiguat in Black obese individuals with insulin resistance. | 12 weeks
  The difference in change in REE between baseline and post-intervention between two arms.

SECONDARY OUTCOMES:
Change in BAT volume after vericiguat in Black obese individuals with insulin resistance. | 12 weeks
  The difference in change in BAT volume between baseline and post-intervention between two arms.
Change in BAT activity after vericiguat in Black obese individuals with insulin resistance. | 12 weeks
  The difference in change in BAT activity between baseline and post-intervention between two arms.
Change in UCP1 gene expression after vericiguat in Black obese individuals with insulin resistance. | 12 weeks
  The difference in change in UCP1 gene expression between baseline and post-intervention between two arms.
Change in exercise energy expenditure (EEE) after vericiguat in Black obese individuals with insulin resistance. | 12 weeks
  The difference in change in EEE between baseline and post-intervention between two arms.
Change in glycosylated hemoglobin (HbA1C) after vericiguat in Black obese individuals with insulin resistance. | 12 weeks
  The difference in change in HbA1C between baseline and post-intervention between two arms.
Change in Body Mass Index (BMI) after vericiguat in Black obese individuals with insulin resistance. | 12 weeks
  The difference in change in BMI between baseline and post-intervention between two arms.
Change in Total Cholesterol (TC) after vericiguat in Black obese individuals with insulin resistance. | 12 weeks
  The difference in change in TC between baseline and post-intervention between two arms.
Change in low-density lipoprotein-cholesterol (LDL-C) after vericiguat in Black obese individuals with insulin resistance. | 12 weeks
  The difference in change in LDL-C between baseline and post-intervention between two arms.

CONTACTS AND LOCATIONS:
Overall Officials: Pankaj Arora, MD, FAHA, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Undecided